CLINICAL TRIAL: NCT06574815
Title: Evaluation of the Effects of the Small Intestine Submucosa (SIS) Biological Membrane on Guided Bone Regeneration (GBR) and Early Loading of Dental Implants in the Maxillary Anterior Region
Brief Title: Effects of the SIS Membrane on GBR and Early Loading of Maxillary Anterior Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Stomatological Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Chao Liang, Doctor of Department of Dental Implant Center, Beijing Stomatological Hospital, Capital Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CMUSH-IRB-KJ-PJ-2023-24; CSA-SIS2022-17 (Other Grant/Funding Number: the Chinese Stomatological Association)
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Dental Implantation; Guided Bone Regeneration
Keywords: Dental implantation; Guided bone regeneration; Early loading; Small intestine submucosa membranes; Randomized controlled trial
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SIS-EL (Experimental): Guided bone regeneration (GBR) with an SIS membrane and early implant loading
  Interventions: Procedure: Early implant loading; Procedure: GBR using an SIS membrane
- Gide-EL (Active Comparator): Guided bone regeneration (GBR) with a Bio-Gide membrane and early implant loading
  Interventions: Procedure: Early implant loading; Procedure: GBR using an Bio-Gide membrane
- Gide-DL (Sham Comparator): Guided bone regeneration (GBR) with a Bio-Gide membrane and delayed implant loading
  Interventions: Procedure: Delayed implant loading; Procedure: GBR using an Bio-Gide membrane

INTERVENTIONS:
Procedure: Early implant loading — Patients underwent definitive restoration at 6 weeks after implant surgery (early loading).
  Arms: Gide-EL; SIS-EL
Procedure: Delayed implant loading — Patients underwent definitive restoration at 6 months after implant surgery (delayed loading).
  Arms: Gide-DL
Procedure: GBR using an SIS membrane — An small intestine submucosa (SIS) membrane was used in the guided bone regeneration (GBR) surgery.
  Arms: SIS-EL
Procedure: GBR using an Bio-Gide membrane — An Bio-Gide membrane was used in the guided bone regeneration (GBR) surgery.
  Arms: Gide-DL; Gide-EL

SUMMARY:
The aim of this randomized controlled trial (RCT) is to determine whether early implant loading that shortens the healing period to 6 weeks can be safely and effectively applied to implants with good initial stability in the maxillary anterior region, which undergoes simultaneous guided bone regeneration (GBR), via clinical examination, intraoral scanning, imageological diagnosis, and aesthetic scoring, and to determine the clinical effect of the small intestine submucosa (SIS) biological barrier membrane in such cases involving early loading. This study is expected to provide preliminary guidance on the timing of loading for a single maxillary anterior implant with insufficient bone volume and provide a theoretical basis for the selection of a biological barrier membrane for GBR in such patients.

DETAILED DESCRIPTION:
Patients were randomized into three groups at a 1:1:1 ratio, including the GBR with a Bio-Gide membrane and delayed implant loading (Gide-DL) group, the GBR with a Bio-Gide membrane and early implant loading (Gide-EL) group, and the GBR with an SIS membrane and early implant loading (SIS-EL) group. The allocation sequence was generated through an online tool (www. random.org) and was concealed in sealed envelopes. At 6 weeks after implant and GBR surgery, the implant stability quotient (ISQ) was measured and recorded at the labial, palatal, mesial, and distal locations via the Osstell device in the Gide-EL group and the SIS-EL group. If the ISQ was ≥ 65, definitive restoration (early loading) was performed (if < 65, the subject was withdrawn from the trial). The digital impressions and occlusal relationships were obtained via intraoral scanning, and the implant-supported crown was designed based on the digital model. Titanium base abutments with angled screw channels (ASCs) and porcelain veneered zirconia (PVZ) crowns were used for restoration. Immediately after definitive restoration, intraoral scanning was used to record the soft tissue contour at the implant site, and CBCT was used to examine the bone tissue around the implant. In addition, patients in the Gide-DL group underwent definitive restoration at 6 months after surgery (delayed loading), and the treatment process was the same as that in the Gide-EL and SIS-EL groups at 6 weeks after surgery. Clinical examination, intraoral scanning, imageological diagnosis, and aesthetic scoring were used to determine the clinical effect of SIS membranes and early implant loading at 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients with single maxillary anterior tooth loss (sites: 12, 11, 21, 22);
* age ≥18 years;
* sex not limited;
* no history of systemic diseases such as heart disease, hypertension, or diabetes;
* no periodontal disease or already received periodontal systemic treatment;
* cone-beam computed tomography (CBCT) revealed that the thickness of the alveolar ridge in the tooth loss area was greater than 3 mm but less than 5 mm;
* using hydrophilic-modified sandblasted and acid-etched (SLActive) bone level tapered (BLT) dental implant systems.

Exclusion Criteria:

* patients receiving radiotherapy and chemotherapy;
* patients with a history of hepatitis, tuberculosis, or other infectious diseases;
* patients with very poor oral hygiene;
* patients who were heavy smokers;
* pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Soft tissue contour assessment | At the 1-year follow-up
  Intraoral scanning was used to collect the soft tissue contour at the implant site, the contour of the implant-supported crown and adjacent natural teeth. The preoperative, immediate postoperative, and 1-year follow-up intraoral scanning data in stereolithography (STL) formats were imported into Exocad 3.0 software. The best-fit images of the median sagittal section at the implant site were extracted, and the horizontal contour changes (HCCs) were measured at 1 mm and 3 mm below the crown-gingiva margin. The preoperative contour was used as the baseline to detect the immediate postoperative horizontal contour increase (HCI), and the immediate postoperative contour was used as another baseline to detect the 1-year follow-up horizontal contour decrease (HCD).
Marginal bone level assessment | At the 1-year follow-up
  X-ray images immediately postoperative (baseline) and at the 1-year follow-up were taken, and the distances from the most coronal bone-to-implant or bone-to-superstructure contact point to the reference point (neck margin of the implant) were measured at the mesial and distal sides of the implant; then, the data were averaged. Negative values were recorded when the contact point was at the root side of the reference point, and positive values were recorded when the contact point was at the crown side of the reference point. The data were calibrated with the known length of the implant to correct for distortion. The MBL changes were obtained by subtracting the baseline data from the 1-year follow-up data.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Liang, PhD, Study Director — Beijing Stomatological Hospital, Capital Medical University
Locations (1):
- Beijing Stomatological Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu R, Yang Z, Tan J, Chen L, Liu H, Yang J. Immediate implant placement for a single anterior maxillary tooth with a facial bone wall defect: A prospective clinical study with a one-year follow-up period. Clin Implant Dent Relat Res. 2019 Dec;21(6):1164-1174. doi: 10.1111/cid.12854. Epub 2019 Nov 11. PMID 31709704
- [Background] Benic GI, Ge Y, Gallucci GO, Jung RE, Schneider D, Hammerle CH. Guided bone regeneration and abutment connection augment the buccal soft tissue contour: 3-year results of a prospective comparative clinical study. Clin Oral Implants Res. 2017 Feb;28(2):219-225. doi: 10.1111/clr.12786. Epub 2016 Feb 8. PMID 26856399
- [Background] Pirc M, Harbeck O, Sapata VM, Husler J, Jung RE, Hammerle CHF, Thoma DS. Contour changes of peri-implant tissues are minimal and similar for a one- and a two-piece implant system over 12 years. Clin Oral Investig. 2021 Feb;25(2):719-727. doi: 10.1007/s00784-020-03638-1. Epub 2020 Oct 15. PMID 33063219
- [Background] Liu Z, Yu X, Ma B, Yang Y, Mu Y, Lu X, Li M, Jing W, Wei P, Ma S, Zhao B, Deng J. SIS membrane modification to improve antimicrobial and osteogenic properties for guide bone regeneration. J Biomater Sci Polym Ed. 2023 Aug;34(10):1337-1359. doi: 10.1080/09205063.2023.2166337. Epub 2023 Jan 17. PMID 36607605
- [Background] Liu Z, Wei P, Cui Q, Mu Y, Zhao Y, Deng J, Zhi M, Wu Y, Jing W, Liu X, Zhao J, Zhao B. Guided bone regeneration with extracellular matrix scaffold of small intestinal submucosa membrane. J Biomater Appl. 2022 Nov;37(5):805-813. doi: 10.1177/08853282221114450. Epub 2022 Aug 4. PMID 35924456
- [Background] Qian SJ, Pu YP, Zhang XM, Wu XY, Liu BL, Lai HC, Shi JY. Clinical, radiographic, and esthetic evaluation of immediate implant placement with buccal bone dehiscence in the anterior maxilla: A 1-year prospective case series. Clin Implant Dent Relat Res. 2023 Feb;25(1):3-10. doi: 10.1111/cid.13154. Epub 2022 Nov 14. PMID 36373737
- [Background] Cairo F, Nieri M, Cavalcanti R, Landi L, Rupe A, Sforza NM, Pace R, Barbato L. Marginal soft tissue recession after lateral guided bone regeneration at implant site: A long-term study with at least 5 years of loading. Clin Oral Implants Res. 2020 Nov;31(11):1116-1124. doi: 10.1111/clr.13658. Epub 2020 Sep 23. PMID 32875633
- [Background] Dard M, Shiota M, Sanda M, Yajima Y, Sekine H, Kasugai S. A randomized, 12-month controlled trial to evaluate non-inferiority of early compared to conventional loading of modSLA implants in single tooth gaps. Int J Implant Dent. 2016 Dec;2(1):10. doi: 10.1186/s40729-016-0040-8. Epub 2016 Apr 4. PMID 27747702
- [Background] Alshhrani WM, Al Amri MD. Customized CAD-CAM healing abutment for delayed loaded implants. J Prosthet Dent. 2016 Aug;116(2):176-9. doi: 10.1016/j.prosdent.2016.01.024. Epub 2016 Mar 30. PMID 27038526
- [Background] Gan LM, Zhou QR, Zhang Y, Yu YC, Yu ZZ, Sun Y, Li RX, Wu XW, Yang F. Alveolar Bone Morphologic Predictors for Guided Bone Regeneration Outcome in Anterior Maxilla. Int Dent J. 2024 Feb;74(1):102-109. doi: 10.1016/j.identj.2023.07.007. Epub 2023 Sep 14. PMID 37714716
- [Background] ElAskary A, Elfana A, Meabed M, Abd-ElWahab Radi I, Akram M, Fawzy El-Sayed K. Immediate implant placement utilizing vestibular socket therapy versus early implant placement with contour augmentation for rehabilitation of compromised extraction sockets in the esthetic zone: A randomized controlled clinical trial. Clin Implant Dent Relat Res. 2022 Oct;24(5):559-568. doi: 10.1111/cid.13120. Epub 2022 Jul 10. PMID 35811090
- [Background] Zuercher AN, Strauss FJ, Paque PN, Bienz SP, Jung RE, Thoma DS. Randomized controlled pilot study comparing small buccal defects around dental implants treated with a subepithelial connective tissue graft or with guided bone regeneration. Clin Oral Implants Res. 2023 Oct;34(10):1094-1105. doi: 10.1111/clr.14140. Epub 2023 Jul 23. PMID 37483129
- [Background] Basler T, Naenni N, Schneider D, Hammerle CHF, Jung RE, Thoma DS. Randomized controlled clinical study assessing two membranes for guided bone regeneration of peri-implant bone defects: 3-year results. Clin Oral Implants Res. 2018 May;29(5):499-507. doi: 10.1111/clr.13147. Epub 2018 Apr 15. PMID 29656495
- [Background] Naenni N, Stucki L, Husler J, Schneider D, Hammerle CHF, Jung RE, Thoma DS. Implants sites with concomitant bone regeneration using a resorbable or non-resorbable membrane result in stable marginal bone levels and similar profilometric outcomes over 5 years. Clin Oral Implants Res. 2021 Aug;32(8):893-904. doi: 10.1111/clr.13764. Epub 2021 Jun 4. PMID 33977571